CLINICAL TRIAL: NCT04197206
Title: Evaluation of Ultrasound Guided Costotransverse Block in Breast Canser Surgery Patients
Brief Title: Ultrasound Guided Costotransverse Block for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cigli Regional Training Hospital (Other)
Responsible Party: Principal Investigator, Hakan Aygün, Principal Investigator,, Cigli Regional Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTB in Breast surgery
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain
Keywords: ultrasound guided block
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costotransverse block (Experimental): The Costotransverse block will be administrated to this group before induction of anesthesia. An intravenous patient-controlled analgesia device within morphine will be given to the patients postoperatively.
  Interventions: Other: costotransverse block
- Control Group (No Intervention): In this group, patients will receive only multimodal analgesic treatment including patient-controlled analgesia with morphine. No block will be performed.

INTERVENTIONS:
Other: costotransverse block — patient controlled analgesia devices with tramadol
  Other Names: patient controlled analgesia
  Arms: Costotransverse block

SUMMARY:
Costotransverse block is a novel regional anesthesia technique described a few months ago. It's use for breast surgery has been reported by only one case report in the literature. As the investigators have considered that Costotransverse block can be efficacious for providing postoperative analgesia in the breast surgeries, the investigators have implemented the application of this blockade into practice at the clinic. The main purpose of this study is to evaluate the analgesic effect of ultrasound-guided unilateral costotransverse block in breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing breast canser surgery under general anesthesia ASA I-II

Exclusion Criteria:

* patients undergoing breast surgery under paravertebral block and others morbidly obesity ASA III - IV infection of the skin at the site of needle puncture area patients with known allergies to any of the study drugs coagulopathy recent use of analgesic/steroid drugs

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
24 hours morphine consumption | 24 hours
  morphine consumptions for both group will be recorded

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Locations (1):
- Cigli regional research hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aygun H, Thomas DT, Nart A. Ultrasound guided single injection costotransverse block in a breast conserving surgery patient; The first clinical report for novel interfascial block. J Clin Anesth. 2020 May;61:109647. doi: 10.1016/j.jclinane.2019.109647. Epub 2019 Oct 26. No abstract available. PMID 31662230
- [Result] Nielsen MV, Moriggl B, Hoermann R, Nielsen TD, Bendtsen TF, Borglum J. Are single-injection erector spinae plane block and multiple-injection costotransverse block equivalent to thoracic paravertebral block? Acta Anaesthesiol Scand. 2019 Oct;63(9):1231-1238. doi: 10.1111/aas.13424. Epub 2019 Jul 23. PMID 31332775
- [Derived] Aygun H, Kiziloglu I, Ozturk NK, Ocal H, Inal A, Kutlucan L, Gonullu E, Tulgar S. Use of ultrasound guided single shot costotransverse block (intertransverse process) in breast cancer surgery: a prospective, randomized, assessor blinded, controlled clinical trial. BMC Anesthesiol. 2022 Apr 18;22(1):110. doi: 10.1186/s12871-022-01651-3. PMID 35436844